CLINICAL TRIAL: NCT05302557
Title: Efferent Loop Stimulation Previous to Ileostomy Closure. Ileostim Trial.
Acronym: Ileostim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Dr. Jorge Arredondo, MD PhD, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ileostim 1.3
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Ileostomy - Stoma; Ileus; Rectal Cancer; Surgical Complication
MeSH Terms: conditions — Ileus; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): During the two weeks prior to the ileostomy closure procedure, daily stimulation of the efferent loop will be performed by irrigation with 500 ml of physiological saline or 500 ml of warm water, preferably bottled, associated with a nutritional thickener. The patient will be instructed by a stomatotherapy nurse. Stimulation will be performed up to the day before the intervention. Kegel exercises will be suggested.
  Every surgeon will use his or her usual technique for all patients included in the study, regardless of the group assigned in the randomization.
  All patients in both groups will receive the same antibiotic and antithrombotic prophylaxis. No antibiotic administration is expected during the postoperative period, following a Zero Surgical Infection (ZSI) protocol.
  Interventions: Other: Ileostomy stimulation
- Control (No Intervention): Direct standard surgery. Every surgeon will use his or her usual technique for all patients included in the study, regardless of the group assigned in the randomization.
  All patients in both groups will receive the same antibiotic and antithrombotic prophylaxis. No antibiotic administration is expected during the postoperative period, following a Zero Surgical Infection (ZSI) protocol.

INTERVENTIONS:
Other: Ileostomy stimulation — Daily stimulation of the efferent loop will be performed during the two weeks prior to the surgery.
  Arms: Interventional

SUMMARY:
The loop ileostomy is an effective method used to bypass faecal contents and reduce the sequelae of possible anastomotic leakage. I t is most often performed after a low anterior resection indicated for lower-middle rectal cancer. A second operation is required for closure, with a morbidity of about 25%.

Many studies have been completed in order to detect possible risk factors - both patient-related and surgery-related - for complications in ileostomy closure surgery. Currently, there is a lack of research studies focused on the preoperative management of these patients.

Our purpose is to reduce the complication rate by optimizing the preoperative status of the distal ileum and to analyze its impact on the reduction of postoperative ileus.

Main objective: To assess whether efferent loop stimulation two weeks before ileostomy closure decreases the incidence of postoperative paralytic ileus.

DETAILED DESCRIPTION:
The loop ileostomy is an effective method used to bypass faecal contents and reduce the sequelae of possible anastomotic leakage. I t is most often performed after a low anterior resection indicated for lower-middle rectal cancer. A second operation is required for closure, with a morbidity of about 25%. Bowel obstruction is the most common complication following this procedure, with an incidence of up to 29%. There is also a risk of anastomotic leakage, observed in 2% of patients, with a reintervention rate approaching 10%. A recent meta-analysis reported up to 2% mortality after stoma reversal.

There are many structural changes in the mucosa of the small bowel after ileostomy formation, which may contribute to the observed morbidity. The distal end may be atrophied, with pathophysiological changes contributing to a reduction in absorptive function and motility.

CONTROVERSY Many studies have been completed in order to detect possible risk factors - both patient-related and surgery-related - for complications in ileostomy closure surgery. Currently, there is a lack of research studies focused on the preoperative management of these patients.

THE NEED FOR SUCH A STUDY There is a high risk of complications following ileostomy reversal (as high as 20%), including bowel dysfunction, anastomotic leakage, bowel perforation and postoperative ileus. This increases the length of hospital stay and healthcare costs.

Our purpose is to reduce this complication rate by optimizing the preoperative status of the distal ileum and to analyze its impact on the reduction of postoperative ileus.

MAIN PURPOSE (OBJECTIVE/GOAL/ SUBJET/PURPOSE) To assess whether efferent loop stimulation two weeks before ileostomy closure decreases the incidence of postoperative paralytic ileus.

SECUNDARY/SIDE/MINOR To evaluate hospital stay and short- and long-term postoperative complications in both groups. To compare postoperative anal continence in both groups.

INCLUSION CRITERIA Patients over 18 years of age who undergo a scheduled protective ileostomy closure surgery, performed in rectal cancer surgery. All patients will follow a homogeneous protocol for testing the rectal anastomosis prior to closure, based on an opaque enema to rule out the presence of anastomotic leakage. Entry into the study does not affect the other surgical indications, in terms of time to ileostomy closure, type of operation or anaesthesia, or request for additional tests. Elective surgery. Patients who sign the informed consent document.

EXCLUSION CRITERIA Patients undergoing simultaneous abdominal procedures at the time of ileostomy closure. History of protective ileostomy for a pathology other than rectal cancer. History of surgery in the ileal region.

BACKGROUND DATA Age, sex, body mass index (calculated as weight in kilograms divided by height in metres squared), American Society of Anesthesiologists (ASA) status and primary diagnosis. Neoadjuvant RT, neoadjuvant QT, time since end of adjuvant chemotherapy. Comorbidities (hypertension, DM, dyslipidaemia, respiratory pathology, others). Complications of the primary tumour surgery. Baseline analytical parameters: proteins, creatinine, ions, Hb and leukocytes.

SURGICAL DATA Operative time (in minutes), presence of parasternal hernia, time from main surgery to ileostomy closure, mesh placement.

EFFERENT LOOP STIMULATION TECHNIQUE:

During the two weeks prior to the ileostomy closure procedure, daily stimulation of the efferent loop will be performed by irrigation with 500 ml of physiological saline or 500 ml of warm water, preferably bottled, associated with a nutritional thickener (Resource, Nestlé Health-science, 6.4g sachet). The patient will be instructed by a stomatotherapy nurse. Stimulation will be performed up to the day before the intervention. Kegel exercises will be suggested.

SURGICAL TECHNIQUE Every surgeon will use his or her usual technique, with a choice between options A and B, using the same technique for all patients included in the study, regardless of the group assigned in the randomization.

Option A. Mechanical closure:

Peri-ileostomy incision. Ileostomy closure technique: anti-peristaltic L-L anastomosis by linear stapler with triple stapling, with endo-stapler closure of the enterotomy and similar loading. Invagination of the staple line.

Option B. Manual closing Peri-ileostomy incision. Ileostomy closure technique: Manual closure of the enterotomy with monofilament or braided suture, using loose stitches or continuous suture, according to standard technique.

All patients will receive the same antibiotic and antithrombotic prophylaxis. No antibiotic administration is expected during the postoperative period, following a Zero Surgical Infection (ZSI) protocol.

PRIMARY OUTCOMES Presence of paralytic ileus (defined as intolerance to oral food on or after the third postoperative day, in the absence of clinical or radiological signs of obstruction, requiring placement of a nasogastric tube or associated with two of the following: nausea/vomiting, abdominal distention and the absence of flatus).

ADDITIONAL, MINOR, SECONDARY OUTCOMES Secondary outcomes will include length of hospital stay, time to tolerate regular diet, time to first passage of flatus, time to first passage of stool, general morbidity [including anastomotic leak, surgical site infection (superficial, deep, organ space), other complications: urinary tract infection, pneumonia, postoperative acute kidney injury, deep vein thrombosis, pulmonary embolism, small bowel obstruction, myocardial infarction, stroke, reoperation and "other". Mortality and diarrhoea. The severity of surgical complications will be classified according to the Clavien-Dindo scale. Grade of postoperative continence and incidence of anterior resection syndrome. Hospital readmission rate.

LONG-TERM OUTCOMES (6 MONTHS):

Readmission rate. Surgical re-intervention. Eventration.

THE STATISTICAL ANALYSIS A comparative analysis will be performed between the two groups according to prior stimulation of the efferent loop or not.

Categorical samples will be analyzed by means of contingency tables and Chi-square. Continuous variables will be examined by comparing means using Student's t-test and medians with the Mann-Whitney U test. Values of p <0.05 will be considered statistically significant. The SPPS 15.0 Inc. Chicago IL. software was used for this purpose.

Sample size estimation: Assuming an alpha risk of 0.05 and a beta risk of 0.2, in a two-tailed test, it is estimated that 68 patients need to be included in each group to find a statistically significant difference in proportions. A ratio of 0.29 in the control group and 0.1 in the intervention group is considered. A loss of patients of 5% is assumed.

Randomization will be performed in a 1:1 ratio in each hospital using the Sealed Envelope simple randomization service program. The researcher will not know the assigned group at the time of offering the study to the patient.

ETHICAL APPROVAL The study will be pre-approved by the local Research Ethics Committee (IRB). Patients will be informed of the possibility of participation in the study by signing the informed consent before being included. The patient will be able to withdraw his/her consent at any time without this affecting the medical care he/she will receive.

The study will be performed in accordance with the Declaration of Helsinki.

FINANCIAL REPORT No financial compensation for participation in the study is foreseen for either the patient or the research team. This study has not received any financial support.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who undergo a scheduled protective ileostomy closure surgery, performed in rectal cancer surgery. All patients will follow a homogeneous protocol for testing the rectal anastomosis prior to closure, based on an opaque enema to rule out the presence of anastomotic leakage. Entry into the study does not affect the other surgical indications, in terms of time to ileostomy closure, type of operation or anaesthesia, or request for additional tests. Elective surgery. Patients who sign the informed consent document.

Exclusion Criteria:

* Patients undergoing simultaneous abdominal procedures at the time of ileostomy closure. History of protective ileostomy for a pathology other than rectal cancer. History of surgery in the ileal region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-12-09 (Estimated); Study Completion 2024-05-09 (Estimated)

PRIMARY OUTCOMES:
Ileus | 1 month
  Presence of paralytic ileus (defined as intolerance to oral food on or after the third postoperative day, in the absence of clinical or radiological signs of obstruction, requiring placement of a nasogastric tube or associated with two of the following: nausea/vomiting, abdominal distention and the absence of flatus).

SECONDARY OUTCOMES:
Hospital stay | 1 month
  Length of hospital stay
Time to tolerate regular diet | 1 month
  Time to tolerate regular diet
Time to first passage of flatus | 1 month
  Time to first passage of flatus
Time to first passage of stool | 1 month
  Time to first passage of stool
General morbidity | 6 months
  General morbidity [including anastomotic leak, surgical site infection (superficial, deep, organ space), other complications: urinary tract infection, pneumonia, postoperative acute kidney injury, deep vein thrombosis, pulmonary embolism, small bowel obstruction, myocardial infarction, stroke, reoperation and "other".
Postoperative continence | 6 months
  Grade of postoperative continence and incidence of anterior resection syndrome
Hospital readmission | 6 months
  Hospital readmission rate

CONTACTS AND LOCATIONS:
Locations (1):
- Jorge Arredondo, León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blanco N, Oliva I, Tejedor P, Pastor E, Alvarellos A, Pastor C, Baixauli J, Arredondo J. ILEOSTIM trial: a study protocol to evaluate the effectiveness of efferent loop stimulation before ileostomy reversal. Tech Coloproctol. 2023 Dec;27(12):1251-1256. doi: 10.1007/s10151-023-02807-0. Epub 2023 Apr 27. PMID 37106220